CLINICAL TRIAL: NCT02739334
Title: PALS-CATCH Intervention for Obesity Prevention Among At-risk Toddlers
Acronym: ENRICH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Shreela V Sharma, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-15-0293
Record Dates: First submitted 2016-03-24; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ENRICH (Experimental): The intervention will integrate the Play and Learning Strategies (PALS) program, a 10-week home-based parent-centered curriculum designed to facilitate parents' mastery of skills for interacting with their toddler with Coordinated Approach To Child Health (CATCH), a behaviorally-based school health promotion program based on Social Cognitive Theory (SCT) to increase opportunities for healthy eating and activity.
  Interventions: Behavioral: ENRICH
- Control - monthly handouts (Active Comparator): The control group receives monthly handouts (one per month) for 3 months that provides information on various topics including child cognitive and language development and child behaviors as it pertains to 2 and 3 year old children.
  Interventions: Behavioral: Control - monthly handouts

INTERVENTIONS:
Behavioral: ENRICH — The intervention, called ENRICH (Encouraging Nurturing Responsiveness to Improve Child Health), is a 10-week home-based parent-centered curriculum designed to facilitate parents' mastery of skills for interacting with their toddler to increase opportunities for healthy eating and activity. Each weekly session is a 60 minute session implemented by a trained coach.
  Arms: ENRICH
Behavioral: Control - monthly handouts — The control group receives monthly handouts (one per month) for 3 months that provides information on various topics including child cognitive and language development and child behaviors as it pertains to 2 and 3 year old children.
  Arms: Control - monthly handouts

SUMMARY:
The purpose of this study is to learn whether a combination of two research-proven programs, a responsive caregiving parenting program and a childhood obesity prevention program, will have an effect on toddlers' healthy nutrition and physical activity behaviors. Investigators hypothesize that the children participating in the intervention will have significantly lower BMI z-scores, lower intake of sugar sweetened beverages, and increased number of servings of fruits and vegetables, and minutes of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* child is 2 - 3 years at the time of enrollment
* child is >85th percentile for BMI
* ability of the parents to speak and read in English at the 4th grade level
* provide primarily in-home care for the children at the time of enrollment
* child is Medicaid eligible

Exclusion Criteria:

* acute secondary complications of obesity for child (e.g., severe respiratory insufficiency)
* child with endocrine abnormalities
* child with severe obesity (>99.5th BMI percentile)
* children who have participated in an obesity treatment program within the past year
* parent with significant sensory impairments (e.g. deaf, blind)
* parent with BMI >40.0

Ages: 24 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
change in child Body Mass Index | baseline and 10 weeks

SECONDARY OUTCOMES:
change in intake of servings of sugar sweetened beverages for the child as assessed using 24 hour parent-reported recalls | baseline and 10 weeks
  investigators will assess intake of sugar sweetened beverages per day as collected using multiple 24 hour recalls with the parents conducted by trained interviewers.
change in total intake of servings fruits and vegetables for the child as assessed using 24 hour parent-reported recalls | baseline and 10 weeks
  investigators will assess total intake of servings of fruit and vegetable per day as collected using multiple 24 hour recalls with the parents conducted by trained interviewers.
change in daily minutes of physical activity for the child as assessed using accelerometers | baseline and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shreela Sharma, PhD, RD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States